CLINICAL TRIAL: NCT06090838
Title: Balloon Pulmonary Angioplasty in Chronic Thromboembolic Pulmonary Disease Without or With Mild Pulmonary Hypertension
Brief Title: BPA in CTEPD Without PH
Acronym: BALLOON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Trombosestichting Nederland (Unknown)
Responsible Party: Principal Investigator, Josien van Es, MD PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL83240.018.23
Record Dates: First submitted 2023-09-11; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Chronic Thromboembolic Disease

STUDY DESIGN:
Intervention Model Description: RCT with cross-over phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention, BPA (Experimental): Will receive questionnaires, exercise testing and BPA at baseline, follow up with questionnaires and exercise testing will be done at 6,12 and 24 months.
  Interventions: Procedure: Balloon Pulmonary Angioplasty (BPA)
- Control, no BPA (No Intervention): Will receive questionnaires, exercise testing at baseline. Due to the crossover design, they will receive BPA at 6 months. Follow up with questionnaires and exercise testing will be done at 6,12 and 24 months.

INTERVENTIONS:
Procedure: Balloon Pulmonary Angioplasty (BPA) — A balloon pulmonary angioplasty is a minimally invasive intervention procedure to remove blood clots from the pulmonary arteries.
  Arms: Intervention, BPA

SUMMARY:
The goal of this clinical trial is to assess the effect of Balloon Pulmonary Angioplasty (BPA) on quality of life and exercise capacity in patients with chronic tromboembolic pulmonary disease (CTEPD) without pulmonary hypertension (PH).

The main question[s] it aims to answer are:

* What is the effect of BPA on quality of life, measured with the PEmb-QoL-questionnaire, in patients with CTEPD without PH?
* What is the effect of is the effect of BPA on exercise capacity in patients with CTEPD without PH?

This study is a randomised clinical trial with cross-over design. Participants will be randomised in an intervention and a control group. At baseline, questionnaires and exercise tests will be perfomed in all patients. The intervention group will first receive BPA-treatment. After 6 months, all patients will fill in the questionaires and undergo the exercise tests. At this point the control group will also receive BPA-treatment. After 12 months the study outcomes will be measured in all participants with the same questionnaires and exercise tests. The total follow-up is 24 months.

DETAILED DESCRIPTION:
BALLOON-TRIAL is a mono-center, prospective, open-label, randomized clinical trial with PROBE design. By adopting a cross-over part, all patients are eventually offered Balloon Pulmonary Angioplasty (BPA) treatment. In addition, this design allows assessment of several important secondary endpoints, such as the duration of the therapeutic effects of the intervention and the most appropriate timing of the intervention. Finally, this design minimizes the influence of confounding covariates, because each patient serves as his or her own control in the evaluation of several secondary endpoints.

As part of clinical care, persistent dyspnea and functional limitations (NYHA class ≥2) are routinely assessed at least three months after the index PE diagnosis. All symptomatic patients are subjected to routine blood testing including Hb, NT-proBNP and creatinine, resting transthoracic echocardiography, computed tomography pulmonary angiography (CTPA), perfusion imaging and/or pulmonary angiography (< 6 months), cardiopulmonary exercise testing (CPET) using a stationary cycle ergometer, Work Rate cycle Test (CWRT) and pulmonary function tests. Furthermore a right heart catheterization will be preferably performed in all patients.

Rehabilitation seems effective and safe in patients with acute PE and in patients with CTEPH, and can be considered standard of care for patients with chronic tromboembolic pulmonary disease (CTEPD) without pulmonary hypertension (PH). Because deconditioning is a known contributor to exercise intolerance after acute pulmonary embolism, patients need to have followed a rehabilitation program of at least 8 weeks before inclusion. Depending on the local protocol, rehabilitation sessions could be daily or a few times a week. Of note, if exercise tests are performed prior to rehabilitation, they should be repeated thereafter to evaluate the effect of rehabilitation, as part of clinical care. Subsequently, all test results are discussed in a multidisciplinary team of PH experts with specific expertise in CTEPH/CTEPD, including cardiologists, pulmonologists, (intervention) radiologists, cardiothoracic surgeons and vascular medicine specialists. Patients diagnosed with CTEPD with mPAP < 25mmHg and PVR < 3WU and who are eligible for this trial will be asked for informed consent for study participation. Of note, if no right heart catheterization is available at screening, patients can still be randomized and in case of a mPAP > 25mmHg, measured by the first BPA, patients will be excluded from the study. After signing informed consent, all PROMS are collected; all questionnaires are automatically distributed by mail and patients are asked to fill in and return digitally.

Patients will be randomized (ratio 1:1) between BPA versus standard of care, which is conservative treatment without specific intervention. Because recovery of symptoms may also occur spontaneously in CTEPD with PVR < 3, the study is controlled by the non-intervention arm. However, all participants will have the opportunity to undergo BPA by during the cross-over phase of the study. The cross-over will take place six months following randomization and after evaluating the primary and secondary outcomes. After the cross-over, patients subjected to the BPA arm will be followed for six months without any intervention. Vice versa, the other cohort will be subjected to BPA following the exact same treatment protocol. All patients will be followed for 24 months. Patients are asked to complete PROMS at randomisation and after 6, 12 and 24 months follow-up. Physical performance, measured by exercise tests will be assessed, in both study arms 6 and 12 months after randomization (and at least 2 months following the last BPA).

The study is unblinded to investigators and patients, but adjudication of the primary outcome measure and will be completed by a blinded committee.

ELIGIBILITY:
Inclusion Criteria:

* acute pulmonary embolism at least 3 months prior to inclusion and adequately treated
* persistent functional limitations: (New York Heart Association (NYHA) class ≥2)
* persistent radiological perfusion defects: ≥ 3 segmental perfusion defects
* CPET result with:

  1. at least 2 of the following criteria:

     * peak VO2 < 80%;
     * peak O2 pulse < 80% of predicted;
     * V'E/V'CO2 @ nadir > 34;
     * Vd/Vt increasing until peak exercise or peak Vd/Vt > 0;4;
     * gradual drop of SpO2 of ≥ 3%;
  2. these exercise findings cannot be explained otherwise 2. patients completed a pulmonary rehabilitation program of at least 8 weeks no longer than 2 months before randomization.

     3. exercise tests were performed after the pulmonary rehabilitation program 4. age 18-80 years 5. Clinical Frailty Scale (CFS) score < 5 (CFS is a 9-point scale that summarizes the overall level of fitness or frailty of an older adult) 6. written informed consent 7. prior treatment or restart therapeutic dose of anticoagulation treatment before randomization

     Exclusion Criteria:
     1. history of balloon pulmonalis angiography (BPA) or pulmonary endarterectomy
     2. residual thrombi that are not eligible for BPA
     3. major acute or chronic cardiopulmonary comorbidities with an expected impact on survival, exercise capacity and/or gas exchange, e.g. significant coronary heart disease, diastolic/systolic heart failure, pulmonary hypertension (mPAP > 25 mmHg), severe chronic obstructive pulmonary disease (COPD) GOLD class ≥3, interstitial lung disease (ILD), disabling neuromuscular disease, malignancy
     4. inability to undergo exercise tests
     5. contrast allergy
     6. creatinine clearance < 30ml/min
     7. pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
disease specific quality of life | baseline, 6 months, 12 months and 24 months
  Quality of life, measured with PEmb-QoL
  The PEmb-QoL is a questionnaire which comprises 40 items and assesses disease-specific QoL during the previous 4 weeks in 6 dimensions: frequency of complaints, activity of daily life (ADL) limitations, work-related problems, social limitations, intensity of complaints, and emotional complaints. The total score is calculated taking into account the difference in total items. The minimum clinically important difference is 15 point.

SECONDARY OUTCOMES:
Change in max load in cardiopulmonary exercise test | baseline, 6 and 12 months
  load in Watt measured at rest, anaerobic threshold and max capacity
Change in oxygen uptake (VO2) in cardiopulmonary exercise test | baseline, 6 and 12 months
  VO2 measured in mL/min and mL/min/kg at rest, anaerobic threshold and max capacity
Change in O2 pulse in cardiopulmonary exercise test | baseline, 6 and 12 months
  O2 pulse measured in VO2/HR measured in ML at rest, anaerobic threshold and max capacity
Change in oxygen saturation in cardiopulmonary exercise test | baseline, 6 and 12 months
  spO2 measured in %, at rest, anaerobic threshold and max capacity
Change in eqCO2 in exercise capacity in cardiopulmonary exercise test | baseline, 6 and 12 months
  eqCO2 is the minute ventilation (VE) in mL divided by the minute volume of CO2 (VCO2) in ML, the eqCO2 is thus described as the VE/VCO2, ans is measured at rest, anaerobic threshold and max capacity
Change in constant work rate test | baseline, 6 and 12 months
  The constant work rate test is an endurance exercise test, in which the participant cycles at a load that is 75% of the max load as measured in the cardiopulmonary exercise test.
  The time in seconds of sustained exercise in this intensity is the outcome measure

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No